CLINICAL TRIAL: NCT06887686
Title: This Study Complies with the Requirements of the Final Rule (42 CFR Part 11) for Clinical Trials with a Start Date of January 18, 2017, or Later, Including the Registration and Reporting of Results As Per the Applicable Regulations.
Brief Title: The Effect of Wiping and Swaddling Bath Methods Applied in the Neonatal Intensive Care Unit on Neonatal Comfort: a Randomized Controlled Trial
Acronym: WS-Bath RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gamze Gocmen (Other)
Responsible Party: Sponsor-Investigator, Gamze Gocmen, ebe, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/01-19
Record Dates: First submitted 2025-03-16; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Care Neonatal Comfort Swaddled Bathing Wipe Bathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Swaddled Bath Group Wipe Bath Group (Experimental): Swaddled Bath Group:
  In this group, infants are wrapped in a soft towel or blanket to maintain a flexed position and then immersed in warm water at an appropriate temperature. The swaddled bath is designed to reduce stress and pain, especially for premature infants. It promotes relaxation, stabilizes the body temperature, and enhances the infant's comfort by reducing crying. The wrapping creates a secure and calming environment that mimics the comforting sensations of the womb, helping to soothe the infant's physiological and behavioral responses.
  Wipe Bath Group:
  In this group, infants are gently wiped with a cloth soaked in warm water. The wipe bath helps maintain body temperature, but it is less invasive than the swaddled bath and does not have the same calming effects. This method is primarily used for cleaning the baby's skin, while not providing as much relaxation or physiological stabilization as the swaddled bath. Although effective for hygiene purposes, it has a milder imp
  Interventions: Behavioral: Swaddled Bath Intervention Wipe Bath Intervention

INTERVENTIONS:
Behavioral: Swaddled Bath Intervention Wipe Bath Intervention — Swaddled Bath Intervention:
  In the swaddled bath group, infants are gently wrapped in a soft towel or blanket to maintain a flexed position. They are then immersed in warm water at an appropriate temperature to regulate body temperature. This intervention is designed to reduce stress and pain, particularly for premature infants, and helps to relax the baby's muscles, stabilize body temperature, and increase overall comfort. It is expected to show a more significant effect on physiological and behavioral stabilization than less invasive methods.
  Wipe Bath Intervention:
  In the wipe bath group, infants are gently wiped with a cloth soaked in warm water. This method is less invasive than the swaddled bath, aiming to maintain body temperature while providing a milder level of relaxation. The wipe bath is effective for skin cleansing but may not provide the same comfort or stress-reducing effects as the swaddled bath. The expected physiological effects, such as body temperature stabilizatio

SUMMARY:
This study will be conducted as a randomized controlled trial to examine the effects of different bathing methods on neonatal comfort. The study will take place in the Neonatal Intensive Care Unit (NICU) of İzmir Tepecik Training and Research Hospital, with a total sample size of 64 neonates who meet the inclusion criteria.

Neonates born at 37 weeks or later, with stable physiological parameters, and receiving their first bath will be included. Those diagnosed with sepsis, on mechanical ventilation, or with impaired skin integrity will be excluded.

The swaddled bath will be applied to the intervention group, while the wipe bath will be applied to the control group. Neonatal comfort levels will be assessed by a second nurse at 10 and 60 minutes after bathing. Data collection will utilize the COMFORT Neo scale, and statistical analyses will be performed using IBM SPSS. T-tests, ANOVA, and correlation tests will be used to compare the effects of bathing methods on neonatal comfort.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to compare the effects of swaddled bathing and wipe bathing on neonatal comfort in Neonatal Intensive Care Units (NICUs). The study will be conducted in the NICU of İzmir Tepecik Training and Research Hospital, and after obtaining ethical approval, 64 neonates meeting the inclusion criteria will be enrolled.

As part of the study, the swaddled bath will be applied to the intervention group, while the wipe bath will be applied to the control group. The bathing procedures will be carried out by the researcher according to standard protocols. Neonatal comfort levels will be assessed by a second nurse working in the NICU at 10 and 60 minutes after bathing, using the COMFORT Neo scale.

Data Analysis:

Collected data will be analyzed using IBM SPSS Statistical Package Program. Descriptive statistics (mean, percentage, standard deviation) will be calculated, and t-tests, ANOVA, and correlation analysis will be conducted to evaluate differences between the groups.

Ethical Considerations:

Prior to the study, approval will be obtained from the Non-Interventional Research Ethics Committee of İzmir Tepecik Training and Research Hospital. Additionally, parents of the neonates will be provided with detailed information about the study, and informed consent will be obtained.

This study aims to contribute to the standardization of bathing methods in NICUs and to determine the most effective technique for improving neonatal comfort.

ELIGIBILITY:
Inclusion Criteria:

* Born at 37 weeks of gestation or later
* Aged between 2 and 7 days
* Born after 24 hours
* Stable physiological parameters
* Spontaneous respiration
* Birth weight ≥ 2000 grams
* No skin problems that would prevent the administration of swaddle or wipe bath
* Both vaginal and cesarean deliveries are accepted

Exclusion Criteria:

* Using sedative or muscle relaxant medications
* Previously exposed to any bath method
* On mechanical ventilation
* Diagnosed with sepsis
* Within the first 78 hours post-operatively
* Having a central catheter
* Having disrupted skin integrity
* Having cranial hemorrhage
* Major congenital, chromosomal, or neurological anomalies

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Newborn comfort (measured with the KONFOR Neo scale) | Data collection will include comfort assessments at the 10th and 60th minutes after the bath.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Ekşioğlu, Doç. Dr., Principal Investigator — Ege University
Locations (1):
- Izmir Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)